CLINICAL TRIAL: NCT06562114
Title: A Phase 1, Safety, Tolerability, Single-ascending Dose, Multiple-ascending Dose, Food Effect, and Pharmacokinetic Study of TML-6 in Healthy Volunteers
Brief Title: A Phase 1 Safety and Tolerability Study of TML-6 in Healthy and Elderly Volunteers for Alzheimer's Disease Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merry Life Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MELTMLZ20220315
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TML-6 Granules (Experimental): This study consists of 5 parts, Part 1 (SAD): 5 cohorts of subjects are planned to be orally dosed, ranging from 100 mg - 1000 mg.
  Part 2 (Food effect): All subjects in Cohort 2 of Part 1 will constitute Period 1 of Part 2 and will move to Period 2 to receive the same Investigational Product (IP) dose as in Period 1.
  Part 3 (Elderly): One cohort of elderly subjects will receive a single dose of IP. A dose level of IP within the safe range defined in the Part 1 SAD study will be chosen
  Part 4 (MAD): 2 cohorts of subjects are planned to be orally dosed once daily for 7 consecutive days, ranging from 400 mg - 800 mg.
  Part 5 (MAD+Cerebrospinal Fluid, CSF PK): One cohort of elderly subjects will receive orally once daily for 7 consecutive days of IP. The dose level of IP defined in the Part 4 MAD study will be chosen.
  Interventions: Drug: TML-6 Granules
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TML-6 Granules — Administered orally
  Arms: TML-6 Granules
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, single-ascending dose (SAD), multiple-ascending dose (MAD), food effect, and pharmacokinetic (PK) Study of TML-6.

ELIGIBILITY:
Healthy adults: Subject's age is ≥18 years old and ≤55 years old at screening Healthy elderly adults: Subject's age is ≥60 years old and ≤80 years old at screening

Inclusion Criteria:

1. Healthy male and female volunteers
2. For Parts 1, 2, and 4 (Cohorts 1-5 and 7-8): Subject's age is ≥18 years old and ≤55 years old at screening.

   For Parts 3 and 5 (Cohorts 6 and 9): Subject's age is ≥60 years old and ≤80 years old at screening.
3. For Parts 1, 2, and 4 (Cohorts 1-5 and 7-8): Subjects whose body mass index (BMI) at screening is within a range of ≥18.5 kg/m2 and <30.0 kg/m2 For Parts 3 and 5 (Cohorts 6 and 9): Subjects whose BMI <30.0 kg/m2 Note: BMI = Body weight (kg) / [Height (m)]2; Body weight is not less than 50 kg at screening and admission.
4. Subjects who are deemed to be satisfactory health by the investigator through an assessment of their medical history, physical examinations, and routine laboratory tests.
5. Female subjects of child-bearing potential show negative pregnancy test results at screening and admission.
6. Female subjects of child-bearing potential, committing to practicing sexual abstinence or using and continue to use 2 highly effective contraceptives of birth control for at least 30 days prior to screening (that period will extend to 90 days for oral contraceptive use) and for at least 30 days after the last dose of investigational product (IP).

   For a subject to be considered not to be of child-bearing potential, she must have been amenorrheic for at least 12 months with confirmed follicle-stimulating hormone (FSH) level (within postmenopausal range) at screening, or must have had a hysterectomy, a bilateral tubal ligation, and/or a bilateral oophorectomy (as determined by the medical history).

   The male partner of a female study subject with childbearing potential must use a condom and ensure that his partner uses a highly effective contraception as outlined below.

   The highly effective contraception methods include:
   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
   3. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
   4. Combination of the following listed methods (d.1+d.2):

   d.1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception, intrauterine device (IUD), or intrauterine system (IUS).

   d.2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).
7. Subjects must demonstrate willingness to comply with all requirements, instructions and restrictions stated in the protocol, and must provide the written informed consent form after thorough understanding.

   -

Exclusion Criteria:

1. Subjects with any properly diagnosed disease within 30 days prior to the first dose of the IP.
2. Subjects who have a QTcF interval >450 msec (male) or >470 msec (female) (Fridericia's correction) at screening. The assessment may be repeated once during the screening period.
3. Systolic blood pressure (SBP) >140 mmHg or diastolic blood pressure (DBP) >90 mmHg at screening and admission, irrespective of anti-hypertensive medication status for the subject. The assessments may be repeated for confirmation after resting for approximately 10 to 30 minutes.
4. Any laboratory values with the following deviations at screening and admission. The laboratory test may be repeated once during the screening period and Day -1.

   • White blood cell count (WBC) < 3000/μL
   * Hemoglobin < 10 g/dL
   * Platelet count < 100000/μL
   * Creatinine > upper limit of normal (ULN)
   * Alanine Aminotransferase (ALT) > ULN
   * Aspartate Aminotransferase (AST) > ULN
   * Total bilirubin > ULN of the reference range * If agreement is obtained per the investigator's discretion, exceptions may be made for isolated ALT or AST elevation <1.5× ULN and bilirubin values that are above the ULN for subject has an underlying diagnosis of Gilbert's syndrome.
5. Subjects who have been tested positive for the following tests:

   - Human immunodeficiency virus (HIV)

   - Hepatitis B virus (HBV)

   - Hepatitis C virus (HCV)
6. Female subjects who are lactating or with a positive pregnancy test at the screening visit and/or admission.
7. Subjects had a history of substance use disorders according to the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-V) criteria.
8. Subjects with positive urine drug test (including cotinine detection) or positive blood alcohol test at screening and on Day -1 (and on Day 15+ in Cohort 2).
9. Subjects with underlying medical, mental, or psychological conditions that may impede study compliance, or, at the discretion of the investigator, preclude participation in the study.
10. The medical history indicates contraindications or hypersensitivity to the use of test medications [TML-6 or any components of the IP].
11. Subjects took any of the following systemically-absorbed medications in the specified durations:

    - Any medications (excluding vitamins, food supplements, and hormonal contraceptives for birth control) within 14 days prior to the first dose of the IP, unless in the opinion of the investigator and sponsor, the medication will not interfere with the study or compromise subject's safety.

    - Any known enzyme inducers/inhibitors or agents that significantly alter hepatic or renal clearance (e.g., erythromycin, cimetidine, barbiturates, phenothiazine, clarithromycin, troleandomycin, ketoconazole, miconazole, fluconazole, itraconazole) within 30 days prior to the first dose of the IP.
12. Subjects had participated in investigational drug trials and took any investigational drug within 30 days or 5 half-lives, whichever is longer, prior to the first dose of the IP.
13. Subjects had blood loss or blood donation of more than 250 and 500 mL within 60 and 90 days, respectively prior to the first dose of the IP.
14. Subjects who cannot stop caffeine-intake for 48 hours prior to the first study dose and during the entire study period.
15. Subjects who are smokers or former smokers who have used nicotine-containing products within 3 months prior to the first dose of the IP.
16. Unwilling or unable to comply with the lifestyle instructions described in the protocol.
17. Subjects appears to have poor venous access.
18. Subjects have any other condition which, in the opinion of the investigator, precludes the subject's participation in the study.

    Additional exclusion criteria for the healthy adult subjects in Cohorts 1-5 and 7-8:
19. Subjects with a clinically significant hematological, endocrine, cardiovascular, hepatic, renal, gastrointestinal, pulmonary, immunologic, metabolic, urologic disorder, and/or malignancy as judged by the investigator; subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism, and excretion of drugs; subjects who has had any previous gastrointestinal surgery, except appendectomy if performed >90 days prior to the first dose of the IP.

    Additional exclusion criteria for the healthy elderly subjects in Cohorts 6 and 9:
20. Subjects with a clinically significant hematological, endocrine, cardiovascular, hepatic, renal, gastrointestinal, pulmonary, immunologic, metabolic, urologic disorder, and/or malignancy that is not well managed and stable, as judged by the investigator; subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism and excretion of drugs; subjects who has had any previous gastrointestinal surgery, except appendectomy if performed >90 days prior to the first dose of the IP.
21. Subjects with estimated Glomerular Filtration Rate (eGFR, calculated based on Cockcroft-Gault formula) of <60 mL/min/1.73 m2 during screening period. If the eGFR exceeds the limits above, the assessment may be repeated once during the screening period.

    Additional exclusion criteria for the subjects in Cohorts 7-9:
22. If the subject has history of suicidal attempt as an adult or suicide ideation in the past year that resulted in pharmacologic treatment or hospitalization, the subject will be excluded if he/she meets any of the following criteria.

    • Answer of "yes" on items 4 or 5 of the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening if the ideation occurred in the previous 6 months.
    * Answer of "yes" on any item of the Suicidal Behavior section of the C-SSRS, except for the Non-Suicidal Self injurious Behavior if this behavior occurred in the previous 2 years.

    Additional exclusion criteria for the subjects in Cohort 9:
23. The subject with clinically significant abnormal finding in the lumbar X-ray examination that is considered incompatible with lumbar puncture (LP) by the investigator at screening.
24. The subject has had CSF collection performed within 30 days prior to Day -1.
25. The subject has a history of clinically significant back pain and/or injury (e.g., clinically significant degenerative disease, spinal deformity, or spinal surgery) that may predispose to complications or technical difficulty with LP, as judged by the investigator.
26. The subject has developed signs and symptoms of spinal radiculopathy, including lower extremity pain and paresthesias.
27. The subject has evidence or history of significant active bleeding or coagulation disorder or have received drugs that affect coagulation or plate function within 14 days prior to LP procedure.
28. The subject has a local infection at the puncture site.
29. The subject has any focal neurological deficit that might suggest an increase in intracranial pressure.
30. The subject has any abnormal finding on ophthalmological assessment/fundoscopy indicative of raised intracranial pressure (i.e., optic disc swelling/edema, or uncontrolled hypertensive retinopathy).
31. The subject has abnormal coagulation tests (prothrombin time [PT]/international normalized ratio [INR], and partial thromboplastin time [PTT]) at screening. The assessment may be repeated once during the screening period.
32. The subject regularly suffers from moderate-to-severe headaches requiring analgesics.
33. Subject's medical history shows hypersensitivity to the anesthetic, or its derivatives used during CSF collection or any medication used to prepare the area of LP procedure.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Incidence of Serious Adverse Events (SAEs) and treatment-related adverse events | All subjects at each dose level complete the 3-day safety assessments post-dose for part 1-3 study and all subjects at each dose level complete the 8-day safety assessments post the first dose for part 4 & 5 study
  Incidence of SAEs and treatment-related severe AEs

SECONDARY OUTCOMES:
Plasma PK: Maximum Plasma Concentration (Cmax) will be assessed for part 1-5 study | Predose, 0.5, 1, 2, 4, 8, 12, 16, 24, and 48 hours postdose
  Part 1-5 study (plasma PK):
  • Peak plasma concentration (PCmax,) [ng/mL] of TML-6
  Part 2 only:
  Comparative bioavailability analysis in the extent of the peak concentration (PCmax)[ng/mL] of TML-6 under fed or fasting condition
Plasma PK: Area Under the Curve (AUC) will be assessed for part 1-5 study | Predose, 0.5, 1, 2, 4, 8, 12, 16, 24, and 48 hours postdose
  Part 1-5 study (plasma PK):
  The TML-6 plasma concentration-time profile will be established and Area under the concentration-time curve (AUC0→24, AUC0→last, 0→inf, and %AUCextrap)[ng*h/mL] of TML-6
  Part 2 only:
  Comparative bioavailability analysis in the extent of total exposure by area under the curve (AUC0→last and AUC0→inf) [ng*h/mL] of TML-6 under fed or fasting condition
Plasma PK: Time to reach peak plasma concentration (Tmax) will be assessed for part 1-5 study | Predose, 0.5, 1, 2, 4, 8, 12, 16, 24, and 48 hours postdose
  Part 1-5 study (plasma PK):
  • Time to reach peak plasma concentration (Tmax)[hours, or h] of TML-6
  Part 2 only:
  Comparative bioavailability analysis in the extent of the Time to reach peak concentration (Tmax)[hours, or h] of TML-6 under fed or fasting condition
Plasma PK: Terminal half-life (T1/2) will be assessed for part 1-5 study | Predose, 0.5, 1, 2, 4, 8, 12, 16, 24, and 48 hours postdose
  Part 1-5 study (plasma PK):
  • Terminal half-life (T1/2) [hour] of TML-6
  Part 2 only:
  Comparative bioavailability analysis in the extent of Terminal half-life (T1/2) [hour] of TML-6 under fed or fasting condition
Plasma PK: Peak plasma concentration at steady state (Cmax,ss) will be assessed for part 4 and 5 study | predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose; Day 3: predose; Day 4:predose; Day 5:predose; Day 6: predose; Day7: predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose
  Part 4-5 study (plasma PK):
  • Peak plasma concentration at steady state (Cmax,ss)[ng/mL] of TML-6
Plasma PK: Area under the concentration-time curve (AUC0→24,ss and AUC0→τ,ss) will be assessed for part 4 and 5 study | predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose; Day 3: predose; Day 4:predose; Day 5:predose; Day 6: predose; Day7: predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose
  Part 4-5 study (plasma PK):
  • Area under the concentration-time curve at steady state (AUC0→24,ss and AUC0→τ,ss) [ng*h/mL] of TML-6
Plasma PK: Time to reach peak concentration at steady state (Tmax,ss) will be assessed for part 4 and 5 study | predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose; Day 3: predose; Day 4:predose; Day 5:predose; Day 6: predose; Day7: predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose
  Part 4-5 study (plasma PK):
  • Time to reach peak concentration at steady state (Tmax,ss) [hours, or h] of TML-6
Plasma PK: Terminal half-life at steady state (T1/2,ss) will be assessed for part 4 and 5 study | predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose; Day 3: predose; Day 4:predose; Day 5:predose; Day 6: predose; Day7: predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose
  Part 4-5 study (plasma PK):
  • Terminal half-life at steady state (T1/2,ss) [hour] of TML-6
Plasma PK: Accumulation ration (Rac) will be assessed for part 4 and 5 study | predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose; Day 3: predose; Day 4:predose; Day 5:predose; Day 6: predose; Day7: predose, 0.5, 1, 2, 4, 8, 12, 16, and 24 hours postdose
  Part 4-5 study (plasma PK):
  • Accumulation ration (Rac) [unit of ratio] of TML-6
CSF PK: Maximum observed concentration in CSF at steady state (CSF Cmax,ss) will be assessed for part 5 study | on Day 7 (prior to dosing, 0.5, 1, 2, 4, 8, 12, 16 hours after dosing) and Day 8 (24 hours after dosing)
  CSF PK at steady-state (after the final dose)
  • Maximum observed concentration in CSF at steady state (CSF Cmax,ss)[ng/mL] of TML-6
CSF PK: Time to reach peak concentration in CSF at steady state (Tmax,ss) will be assessed for part 5 study | on Day 7 (prior to dosing, 0.5, 1, 2, 4, 8, 12, 16 hours after dosing) and Day 8 (24 hours after dosing)
  CSF PK at steady-state (after the final dose),
  • Time to reach peak concentration in CSF at steady state (Tmax,ss) [hours, or h] of TML-6
CSF PK: Area under the CSF concentration-time curve from 0 to the 24 hours at steady state (CSF AUC0→24,ss) will be assessed for 5 study, if applicable | on Day 7 (prior to dosing, 0.5, 1, 2, 4, 8, 12, 16 hours after dosing) and Day 8 (24 hours after dosing)
  CSF PK at steady-state (after the final dose),
  • Area under the CSF concentration-time curve from 0 to the 24 hours at steady state (CSF AUC0→24,ss)[ng*h/mL] of TML-6, if applicable
CSF PK: Ratio of CSF AUC0→24,ss to Plasma AUC0→24,ss for part 5 study, if applicable | on Day 7 (prior to dosing, 0.5, 1, 2, 4, 8, 12, 16 hours after dosing) and Day 8 (24 hours after dosing)
  • Ratio of CSF AUC0→24,ss to Plasma AUC0→24,ss[unit of ratio] of TML-6, if applicable

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No